CLINICAL TRIAL: NCT03420521
Title: An Open-Label, Single Arm Phase II Study of Nivolumab in Combination With Ipilimumab in Subjects With Advanced Neuroendocrine Tumors
Brief Title: Nivolumab With Ipilimumab in Subjects With Neuroendocrine Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J17156; IRB00151698 (Other: JHM IRB)
Record Dates: First submitted 2017-11-30; First posted 2018-02-05 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Neuroendocrine Tumors; Carcinoid Tumor
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab plus Ipilimumab (Other): Nivolumab 240 mg IV over 60 minutes every 2 weeks (Q2W) Ipilimumab 1mg/kg IV over 30 minutes every 6 weeks (Q6W)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — 240mg IV over 60 minutes Q2W
  Other Names: Bristol Myers Squibb (BMS), BMS-936558
Drug: Ipilimumab — 1mg/kg IV over 30 minutes Q6W
  Other Names: Bristol Myers Squibb (BMS), BMS-734016

SUMMARY:
This is a single arm open-label design study looking at Nivolumab plus Ipilimumab in patients with Advanced Neuroendocrine Tumors. Patients will be dosed Nivolumab 240mg IV over 60 minutes every 2 weeks (Q2W) and Ipilimumab 1mg/kg IV over 30 minutes every 6 weeks (Q6W). One cycle will include 3 doses of Nivolumab and 1 dose of Ipilimumab. The objective of this study is to evaluate the objective response rate of combination Nivolumab and Ipilimumab in advanced, well-differentiated neuroendocrine tumors. Durability of response, and progression free survival (PFS) will also be described.

DETAILED DESCRIPTION:
Subjects with progressive, non-functional advanced or metastatic thoracic, GI or pancreatic well-differentiated neuroendocrine tumors (NET) have few treatment options. The only FDA approved treatment regimen offers little response potential. In currently unpublished data with inhibitory immune checkpoint agents, patients with NET have shown promising clinical benefit. This therapy offers a novel approach to potentially provide long term benefit, but must be further explored. The safety profile of nivolumab plus ipilimumab is characterized by immune-related toxicities, such as diarrhea, rash, pneumonitis, liver toxicity, and endocrinopathies (Nivolumab, Ipilimumab Investigator's Brochures). The frequencies and intensities of these events in the combination are variable and depend on the specific doses and schedule used. In the dosing schedules selected, these events were mostly low grade and manageable with the use of corticosteroids. Nivolumab and ipilimumab combination therapy has shown improved efficacy over either agent alone in melanoma. Rationale for Single Arm Design This study will use a single arm open-label design. The objective of this study is to evaluate the objective response rate of combination nivolumab and ipilimumab in advanced, well-differentiated neuroendocrine tumors. Durability of response, and PFS will also be described.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically confirmed advanced, progressive, well-differentiated nonfunctional NET of the pancreas, lung or gastrointestinal (GI) tract per the 8th International Association for the Study of Lung Cancer classification (IASLC) or the American Joint Committee on Cancer (AJCC) Staging Handbook, 7th edition. Progression must be documented over the prior 12 months.

  * Measurable disease by CT or MRI per RECIST 1.1 criteria (Appendix 3); radiographic tumor assessment performed within 28 days before treatment. Target lesions may be located in a previously irradiated field if there is documented (radiographic) disease progression in that site after the completion of radiation therapy.
  * Prior therapy, including everolimus, octreotide, surgery, chemoradiation, is all permitted after being properly noted. This prior therapy must have been completed at least 28 days prior to study enrollment.
  * Patients with lung NETs must have progressed after at least 1 line of therapy. Patients with GI NETs must have had at least 2 lines of prior therapy.
  * Subjects are to have tumor tissue sample available at central lab for programmed cell death ligand 1 (PD-L1) immunohistochemistry (IHC) testing during the screening period. Subjects can initiate therapy before the result of IHC testing.
  * (Stage 2 only) Subjects must be willing to undergo 2 sets of core needle biopsies (pre-treatment and at 6-8 weeks on therapy) if there are lesions amenable to biopsy. Subjects without a lesion amendable to biopsy will still be permitted to enroll provided they have an archival tumor sample for PD-L1 IHC testing. An optional core biopsy will be requested at progression.
  * Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 (see Appendix 1)
  * Prior palliative radiotherapy to non-central nervous system (CNS) lesions must have been completed at least 2 weeks prior to treatment. Subjects with symptomatic tumor lesions at baseline that may require palliative radiotherapy within 4 weeks of first treatment are strongly encouraged to receive palliative radiotherapy prior to treatment.
  * Patients must have normal organ and marrow function as defined below:
* - white blood cell (WBC) ≥1,500/microliters (mcL)
* - absolute neutrophil count ≥1,000/mcL
* - hemoglobin ≥ 8.0 g/dL
* - platelets ≥75,000/mcL
* - total bilirubin ≤ 1.5 x institutional ULN (patients with Gilbert's syndrome may have serum bilirubin ≤ 3 x ULN)
* - aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 × institutional ULN (≤ 5 x ULN in the presence of liver metastases)

  - creatinine
* ≤ 1.5 × institutional ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):
* Female:
* CrCl = (140 - age in years) x weight in kg x 0.85

  o 72 x serum creatinine in mg/dL
* Male:
* CrCl = (140 - age in years) x weight in kg x 1.00

  - 72 x serum creatinine in mg/dL
  * Age ≥18 years of age
  * Patients must have recovered from adverse events due to prior treatment to ≤ grade 1, except for alopecia and sensory neuropathy ≤ grade 2.
  * Patients must be able to understand and the willingness to sign a written informed consent document.
* Exclusion Criteria:

  * Subjects with poorly differentiated or small cell carcinoma histology
  * Subjects with disease that is amenable to surgical resection.
  * Subjects with history of or active symptoms of carcinoid or hormonal syndromes are permitted if symptoms are controlled with a somatostatin analog.
  * Hepatic intra-arterial embolization or peptide receptor radionuclide therapy (PRRT) within 4-8 weeks; cryoablation, radiofrequency ablation or trans-arterial chemoembolization of hepatic metastases within ≤ 4 weeks of study enrollment
  * Subjects with symptomatic untreated CNS metastases are excluded.
  * Subjects are eligible if CNS metastases are asymptomatic or adequately treated and subjects are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to first treatment.
  * In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of <10 mg daily prednisone (or equivalent) for at least 2 weeks prior to first treatment.
  * Subjects with carcinomatous meningitis
  * Subjects must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before first treatment.
  * Pregnant or breast-feeding women
  * Women of child-bearing potential, who are biologically able to conceive, and not employing two forms of highly effective contraception. Highly effective contraception must be used throughout the trial and up to 8 weeks after the last dose of study drug (e.g. male condom with spermicidal; diaphragm with spermicide; intra-uterine device). Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test ≤ 14 days prior to starting study drug.
  * Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
  * Other active malignancy requiring concurrent intervention.
  * Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first treatment. Inhaled or topical steroids, and adrenal replacement steroid 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
  * Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
  * Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
  * Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interferes with the interpretation of safety results.
  * Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
  * Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
  * History of allergy or hypersensitivity to study drug components

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Hann, MD/PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institution, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab Plus Ipilimumab: Nivolumab 240mg IV over 60 minutes every 2 weeks (Q2W) Ipilimumab 1mg/kg IV over 30 minutes every 6 weeks (Q6W)
  Nivolumab: 240mg IV over 60 minutes Q2W
  Ipilimumab: 1mg/kg IV over 30 minutes Q6W
Period: Overall Study
Arm/Group | Nivolumab Plus Ipilimumab
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Nivolumab Plus Ipilimumab: Nivolumab-240 mg IV over 60 minutes Q2W Ipilimumab 1mg/kg IV over 30 minutes Q6W
  Nivolumab: 240mg IV over 60 minutes Q2W
  Ipilimumab: 1mg/kg IV over 30 minutes Q6W
Arm/Group | Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9
Tumor Site [Count of Participants; unit: Participants] — Location of tumor in the body
  Participants
    Lung | 6
    Pancreatic Neuroendocrine | 2
    Small Bowel | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) of Neuroendocrine Tumor (NET) of the Lung, Pancreas, and Gastrointestinal (GI) Tract
Description: The number of subjects who have at least one scan with an Objective Response (OR) of confirmed complete response (CR) or partial response (PR), per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions as assessed by CT scan: Objective Response (OR), a response of CR or PR from baseline to PD, palliative local therapy, or subsequent anticancer therapy; Complete Response (CR), the disappearance of all target lesions and any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm; Partial Response (PR), >= 30% decrease in the sum of the longest diameters of target lesions, compared to baseline sum diameters
Time Frame: up to 24 months
Population: One patient passed away during cycle 1 of therapy, from unrelated issue (colitis, not related to study drug) prior to first RECIST scans, thus was not assessable for ORR, DCR or DOR.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 8
Participants | 4

2. Secondary Outcome: Number of Patients Experiencing Drug-related Adverse Events
Description: Safety as assessed by number of patients experiencing drug-related adverse events (safety and tolerability).
Time Frame: up to 27 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 9
Participants | 8

3. Secondary Outcome: Number of Patients Experiencing Dose-limiting Toxicities
Description: Safety as assessed by number of patients experiencing dose-limiting toxicities (safety and tolerability).
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 9
Participants | 2

4. Secondary Outcome: Progression Free Survival (PFS) at 6 Months
Description: Percentage of patients treated with nivolumab and ipilimumab with no progressive disease (PD) at 6 months using Kaplan Meier estimate, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT scan: Progressive Disease (PD), >= 20% increase in sum of target lesions' diameters, compared to smallest sum on study (including baseline sum, if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of new lesions.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 9
percentage of participants | 44

5. Secondary Outcome: Progression Free Survival (PFS) at 12 Months
Description: Percentage of patients treated with nivolumab and ipilimumab with no progressive disease (PD) at 12 months using Kaplan Meier estimate, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT scan: Progressive Disease (PD), >= 20% increase in sum of target lesions' diameters, compared to smallest sum on study (including baseline sum, if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of new lesions.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 9
percentage of participants | 44

6. Secondary Outcome: Progression Free Survival (PFS) at 24 Months
Description: Percentage of patients treated with nivolumab and ipilimumab with no progressive disease (PD) at 24 months using Kaplan Meier estimate, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT scan: Progressive Disease (PD), >= 20% increase in sum of target lesions' diameters, compared to smallest sum on study (including baseline sum, if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of new lesions.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 9
percentage of participants | 33

7. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Time (months) from date of randomization to progressive disease (PD) or death, whichever comes first, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT scan: Progressive Disease (PD), >= 20% increase in sum of target lesions' diameters, compared to smallest sum on study (including baseline sum, if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of new lesions.
Time Frame: approximately 3 years 8 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 9
months | 5.29 [2.7 to NA] — estimation has not been reached

8. Secondary Outcome: Efficacy as Assessed by Disease Control Rate (DCR)
Description: The number of subjects who have at least one scan with best overall response (BOR) of confirmed complete response (CR), partial response (PR), or stable disease (SD), per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions as assessed by CT scan: Best Overall Response (BOR), best response (CR, PR, or SD) from baseline to PD, palliative local therapy, or subsequent anticancer therapy; Complete Response (CR), the disappearance of all target lesions and any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm; Partial Response (PR), >= 30% decrease in the sum of the longest diameters of target lesions, compared to baseline sum diameters; Stable Disease (SD), <20% increase, <30% decrease in the sum of the longest diameter of target lesions, no measurable increase in non-target lesions, and no new lesions.
Time Frame: approximately 3 years 8 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 8
Participants | 4

9. Secondary Outcome: Efficacy as Assessed by Duration of Response (DOR)
Description: Time (months) from best overall response (BOR) of complete response (CR) or partial response (PR) to progressive disease (PD), per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions by CT scan: Best Overall Response (BOR), best response (CR, PR, or SD) from baseline to PD, palliative local therapy, or subsequent anticancer therapy; Complete Response (CR), the disappearance of all target lesions and any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm; Partial Response (PR), >= 30% decrease in the sum of the longest diameters of target lesions, compared to baseline sum diameters; Progressive Disease (PD), >= 20% increase in sum of target lesions' diameters, compared to smallest sum on study (including baseline sum, if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of new lesions.
Time Frame: approximately 3 years 8 months
Population: The duration of response is in reference to those patients who have had an objective response. In our study, 4 patients had an objective response, thus we reported duration of response on those 4 patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 4
months | NA [8.51 to NA] — estimation has not been reached

10. Secondary Outcome: Efficacy as Assessed by Overall Survival (OS)
Description: Number of months participants stay alive after treatment with the combination of nivolumab and ipilimumab in subjects with advanced well-differentiated nonfunctional NET of the lung, pancreas or GI tract
Time Frame: approximately 3 years 8 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 9
months | NA [19.12 to NA] — estimation has not been reached

ADVERSE EVENTS:
Time Frame: approximately 3 years 8 months
Arm/Group | Nivolumab Plus Ipilimumab
All-Cause Mortality (participants affected / at risk) | 4/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab Plus Ipilimumab (N=9)
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab Plus Ipilimumab (N=9)
Anemia (Blood and lymphatic system disorders) | 5 (7)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (3)
Hypothyroidism (Endocrine disorders) | 3 (7)
Blurred vision (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Eye duct inflammation (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (16)
Anal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (5)
Diarrhea (Gastrointestinal disorders) | 6 (22)
Dry mouth (Gastrointestinal disorders) | 1 (2)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 8 (12)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5)
Chills (General disorders) | 1 (1)
Edema face (General disorders) | 3 (4)
Edema limbs (General disorders) | 3 (8)
Edema neck (General disorders) | 1 (1)
Edema periorbital (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (2)
Fatigue (General disorders) | 7 (21)
Fever (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2)
Upper respiratory infection (Infections and infestations) | 2 (3)
Bruising (Injury, poisoning and procedural complications) | 2 (5)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (10)
ALT increased (Investigations) | 3 (5)
AST increased (Investigations) | 2 (3)
BUN increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 3 (6)
HbA1c increased (Investigations) | 1 (1)
Lactate dehydrogenase increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 2 (23)
Lymphocyte count decreased (Investigations) | 4 (14)
Serum amylase increased (Investigations) | 1 (18)
Weight loss (Investigations) | 2 (4)
Acidosis (Metabolism and nutrition disorders) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5)
Baker's cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1)
Nipple sensitivity (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 3 (4)
Urinary urgency (Renal and urinary disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (4)
Peeling skin on hands (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (10)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (19)
Flushing (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT03420521/Prot_SAP_000.pdf